CLINICAL TRIAL: NCT01818050
Title: Prospective Evaluation of Stent Patency in Patients With Benign Biliary Obstruction of the Wing Biliary Stent (Viaduct™)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: GI Supply (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21604
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Bile Duct Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Wing stent arm (Other): There is only one arm in this study. Intervention: checking liver function tests to evaluate stent patency
  Interventions: Other: Liver Function Tests

INTERVENTIONS:
Other: Liver Function Tests — LFTs will be checked periodically after Wing stent placement to evaluate stent patency

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) with plastic stent placement for resolution of biliary obstruction has been the method of choice for many years. However, stent clogging/obstruction is a major limitation in the management of biliary obstruction. Studies have shown that the conventional tubular type polyethylene stents (CS) with side holes accumulate significant sludge and their mean patency is approximately 90 days.

Thus patients requiring longer term stenting need to undergo stent exchanges every 2-3 months.

Recently, a stent with a star-shaped cross-section has been developed for biliary applications. This FDA approved biliary Wing stent (WS) (ViaDuct™) is a novel plastic biliary stent that lacks a lumen, and is designed to allow bile to flow on the outside of the stent. The stent which is star shaped in cross section, channels fluid along its winged perimeter. It has been proposed that the winged stent design with a lack of central lumen obviates the risk of luminal occlusion and that the risk of occlusion, given the presence of multiple external drainage channels, is smaller. Longer term biliary drainage without the need for stent exchange should therefore be possible with these stents.

The primary aim of this study is to prospectively evaluate the patency rate of the WS up to 90 days in 50 patients with biliary obstruction due to stones or benign strictures.

DETAILED DESCRIPTION:
1. Fifty patients that meet all the inclusion criteria and have none of the exclusion criteria will be invited to participate in the study.
2. Initial visit:

   * Written informed consent will be obtained
   * Complete history and physical will be performed and the patients baseline liver function tests and imaging results will be assessed and noted in the case report form.
   * Patients gender, date of birth, concomitant medications will be noted.
3. Procedure:

   Patients will then be scheduled for the ERCP procedure with wing biliary stent placement. They will undergo the ERCP as standard of care and the wing biliary stent will be placed for decompression of the obstructed biliary system in situations where stenting is standard of care. One or more biliary stents may be placed during the procedure depending on the indication such as a biliary stricture necessitating multiple stent placements for dilation as the standard of care.
4. Bloodwork:

   Patients will undergo bloodwork (total and direct bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase) one week after the procedure. The degree of drop in bilirubin will also be noted. The patients will be then have these labs drawn again at 4, 8 and 12 weeks after the procedure.
5. Telephone calls:

   The patients will be called on the telephone at weeks 2, 4, 6, 8, 10 after the procedure to monitor their clinical status. Patients and family members will be given a contact number to call us immediately if they develop any signs of biliary obstruction such as fever, abdominal pain, jaundice, dark urine or light stools. They will also be instructed to come to the emergency room should they develop fevers.
6. Stent removal:

   At the end of 90 days from the stent placement patients will return for a repeat ERCP for stent removal as the standard of care and further endo-therapy as indicated.
7. Stent patency will be calculated from the time of stent insertion up to the end of 90 days. The stent patency rate at 90 days will be the proportion of stents placed that do not occlude over this time period. Stent occlusion will be defined as biochemical or clinical evidence of obstructive jaundice.
8. All the continuous and outcome variables (stent obstruction) will be statistically analyzed and stent malfunction rates will be analyzed for the wing stent across the various indications.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 or older referred for ERCP for biliary obstruction from stones or benign strictures that have been confirmed based on clinical, laboratory and imaging findings, with an indication for plastic stent placement.

One or more biliary stents may be placed during the procedure depending on the indication such as a biliary stricture necessitating multiple stent placements for dilation as the standard of care.

* Expected patient survival of at least 90 days
* High likelihood of patient follow-up
* Patient is able to give a written informed consent
* Patient is willing and able to comply with the study procedures.

Exclusion Criteria:

* Patients with cholangitis
* Patients with bile leak
* Pregnant patients
* Patients with any contraindication to endoscopic procedure
* Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit
* Patients with malignant biliary strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Biliary stent patency | At 90 days after stent placement

SECONDARY OUTCOMES:
Liver Function Test improvement | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Subhas Banerjee, Principal Investigator — Stanford University; Rajan Kochar, MD, Study Director — Stanford University
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

REFERENCES:
- [Derived] Schmidt A, Riecken B, Rische S, Klinger C, Jakobs R, Bechtler M, Kahler G, Dormann A, Caca K. Wing-shaped plastic stents vs. self-expandable metal stents for palliative drainage of malignant distal biliary obstruction: a randomized multicenter study. Endoscopy. 2015 May;47(5):430-6. doi: 10.1055/s-0034-1391232. Epub 2015 Jan 15. PMID 25590188